CLINICAL TRIAL: NCT01542099
Title: The Effect Site Concentration of Remifentanil Blunting Hemodynamic Responses to Tracheal Intubation: Single Versus Double Lumen Tube
Brief Title: The EC50 of Remifentanil Blunting Hemodynamic Response to Double Lumen Tube Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JHBahk_DLT_remi
Record Dates: First submitted 2012-02-09; First posted 2012-03-02 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Hemodynamic Responses During Tracheal Intubation
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single lumen tube (Active Comparator): Single lumen tube intubation during remifentanil infusion
  Interventions: Drug: Remifentanil
- Double lumen tube (Active Comparator): Double lumen tube intubation during remifentanil infusion
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — According to previous patient's response, the investigators will allocate the effect site concentration of remifentanil of next patient during double lumen tube intubation. For this allocation of dose of remifentanil the investigators use up-and-down method.
  For the first patient, the dose of remifentanil would be fixed at 6.0 ng/ml which we predict as EC50. And, step size of dose is 0.5ng/ml.
  Arms: Double lumen tube
Drug: Remifentanil — According to previous patient's response, the investigators will allocate the effect site concentration of remifentanil of next patient during single lumen tube intubation. For this allocation of dose of remifentanil the investigators use up-and-down method.
  For the first patient, the dose of remifentanil would be fixed at 6.0 ng/ml which we predict as EC50. Step size of dose is 0.5ng/ml.
  Arms: Single lumen tube

SUMMARY:
The purpose of this study is to evaluate the effect site concentration of remifentanil blunting hemodynamic changes to tracheal intubation of single or double lumen tubes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery that require one lung ventilation

Exclusion Criteria:

* patient who does not agree with this study
* BMI < 16.0 or BMI > 30
* cardiovascular disease, pulmonary disease, renal disease
* alcoholic abuser or drug abuser
* patient who takes any drug to influence cardiovascular system or sympathetic nervous system
* any use of local anesthetics or drugs to influence cardiovascular system during tracheal intubation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in heart rate and mean arterial pressure after intubation | intubation period
  Heart rate and mean arterial pressure will be recorded at 2 minutes before intubation, 1 minute before intubation, during intubation, 1 minute after intubation. The mean value of heart rate and mean arterial pressure before intubation will be regarded as the baseline values. If maximum heart rate or mean arterial pressure after intubation increased by >15% from baseline value, the response will be regarded as "fail" and increased concentration of remifentanil will be applied to next patient by up and down sequential method.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim TK, Hong DM, Lee SH, Paik H, Min SH, Seo JH, Jung CW, Bahk JH. Effect-site concentration of remifentanil required to blunt haemodynamic responses during tracheal intubation: A randomized comparison between single- and double-lumen tubes. J Int Med Res. 2018 Jan;46(1):430-439. doi: 10.1177/0300060517721072. Epub 2017 Jul 21. PMID 28730932